CLINICAL TRIAL: NCT04809038
Title: Dry Needling Versus Magnesium Sulphate Iontophoresis in Chronic Mechanical Neck Pain
Brief Title: Dry Needling Versus Magnesium Sulphate Iontophoresis in Subjects With Chronic Mechanical Neck Pain
Acronym: DN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, al shaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p.t.REC/012/003108
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
Keywords: dry needling, iontophoresis, neck pain
MeSH Terms: conditions — Chronic Pain; Neck Pain | interventions — Dry Needling; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: this trial has three group; two experimental and one control
Who Masked: Participant
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dry needling (Experimental): dry needling will be received twice a week for four weeks
  Interventions: Other: dry needling; Other: stretching exercise
- magnesium sulphate iontophoresis (Experimental): magnesium sulphate iontophoresis will be received twice a week for four weeks
  Interventions: Other: magnesium sulphate iontophoresis; Other: stretching exercise
- stretching exercise (Active Comparator): stretching will be received twice a week for four weeks
  Interventions: Other: stretching exercise

INTERVENTIONS:
Other: dry needling — Patient will be placed in a comfortable prone position and encouraged to maintain complete relaxation. The selected active MTrPs was prepared by wiping the area with alcohol pad, and a gauge needle with its plastic guide tube in place will be palced over the active MTrPs .a tapping motion will be used to advance the needle to a depth of 5 to 10 mm for 30 seconds
  Arms: dry needling
Other: magnesium sulphate iontophoresis — The subjects in the iontophoresis group received MgSO4 iontophoresis using an iontophoretic drug delivery system (Phoresor_IIAuto,ModelPM850,IOMED. MTrPs were examined using pincer palpation and marked by pin. MgSO4 was applied to the active positive electrode using a syringe with a concentration of 100 mg/cm2. The active electrode was placed directly over the marked area where the sensitive MTrPs were located. The dispersive electrode was applied to the skin 6 inches distal from the active electrode.
  Arms: magnesium sulphate iontophoresis
Other: stretching exercise — The patient will be placed in a comfortable and relaxed sitting position with his back supported ; one hand was placed on the side of the head applying the stretching force, while the other hand was placed on the patients shoulder applying shoulder stablization . The direction of stretched force was in flexion , side bending to the opposite side and rotation to the same side . The stretched position will be sustained for 30 seconds , then a relaxation period of 30 seconds . This procedure was repeated 3 times .

SUMMARY:
the aim of this trial is to compare dry needling and magnesium sulphate iontophoresis in subjects with mechanical neck pain

DETAILED DESCRIPTION:
Mechanical neck pain is a prevalent condition in various populations. Neck pain occurrence is affected by several factors, involving environmental, psychological, and social aspects. Neck pain represents the fourth major disorder responsible for a person's year lived with disability and ranked eleventh as disability-adjusted life years of a person. The neck pain incidence ranges from 10.4 to 23.3% in 1-year time, while the range of prevalence was 0.4 to 86.8%. It has a high prevalence among computer users, office workers, and females, especially females aged 35 to 49 years old. Myofascial trigger point (MTrP) might play an important role in the formation of mechanical neck pain and is known as a hyperirritable spot in skeletal muscle that is accompanied with a hypersensitive palpable nodule in a taut band.

dry needling and iontophoresis play a major role in the treatment of mechanical neck pain so this trial was conducted to determine which one has superiority. this trial has three groups. two experimental and one control group.pain, function, pressure pain threshold and emg will be measured

ELIGIBILITY:
Inclusion Criteria:

All patients had active trigger myofascial trigger points (MTrPs) in upper trapeziues muscle in the dominant side with mechanical neck pain.

The patients age ranged from 18-35years The patients had been choosen from both sexes . patient agrees not to receive additional treatment for their painful condition during the trial (apart from NSAIDs and pain killers The patients body mass index < 30 kg/m²

Exclusion Criteria:

History of whiplash injury History of cervical spine surgery Cervical radiculopathy or myelopathy Having undergone physical therapy within the past 3 months before the study. Non -rheumatologic diseases as multiple sclerosis , thyroid dysfunction and chronic infection

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  pain will be measured by visual analogue scale
muscle activity in the form of normalized root mean square | up to four weeks
  muscle activity will be measured by electromyograph

SECONDARY OUTCOMES:
function | up to four weeks
  neck function will be measured by Arabic neck disability index
pressure pain threshold | up to four weeks
  pressure pain threshold will be measured by pressure algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shaymaa Shaaban Abd El Azeim, Giza, Egypt